CLINICAL TRIAL: NCT02395172
Title: A Phase III Open-Label, Multicenter Trial of Avelumab (MSB0010718C) Versus Docetaxel in Subjects With Non-Small Cell Lung Cancer That Has Progressed After a Platinum-Containing Doublet
Brief Title: Avelumab in Non-Small Cell Lung Cancer (JAVELIN Lung 200)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100070-004; 2014-005060-15 (EudraCT Number)
Record Dates: First submitted 2015-02-27; First posted 2015-03-20 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Avelumab; MSB0010718C; Non-Small Cell Lung Cancer; Anti-PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avelumab (Experimental)
  Interventions: Drug: Avelumab
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Avelumab — Participants received 10 milligrams per kilogram (mg/kg) of avelumab as a 1-hour intravenous infusion once every 2 weeks until confirmed disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or Investigational Medicinal Product (IMP) as defined in the study protocol was fulfilled.
  Arms: Avelumab
Drug: Docetaxel — Participants received 75 mg per square meter (m^2) (per label) of docetaxel by intravenous infusion once every 3 weeks until confirmed disease progression, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the study or Investigational Medicinal Product (IMP) as defined in the study protocol was fulfilled.
  Arms: Docetaxel

SUMMARY:
The main purpose of this study was to demonstrate superiority with regard to overall survival of avelumab versus docetaxel in participants with programmed death ligand 1 (PD-L1) positive, non-small cell lung cancer (NSCLC) after failure of a platinum-based doublet.

ELIGIBILITY:
Inclusion Criteria

* Signed written informed consent before any trial related procedure
* Male or female participants aged greater than or equal to (>=) 18 years
* Availability of a formalin-fixed, paraffin-embedded block containing tumor tissue or 7 unstained tumor slides suitable for PD-L1 expression assessment
* Tumor determined to be evaluable for PD-L1 expression per the evaluation of a central laboratory
* Participants with histologically confirmed Stage IIIb/IV or recurrent NSCLC who have experienced disease progression
* Participants must have progressed after an acceptable therapy defined as follows:

  1. Participants must have progressed during or after a minimum of 2 cycles of 1 course of a platinum based combination therapy administered for the treatment of a metastatic disease. A history of continuation (use of a non platinum agent from initial combination) or switch (use of a different agent) maintenance therapy is permitted provided there was no progression after the initial combination. A switch of agents during treatment for the management of toxicities is also permitted provided there was no progression after the initial combination OR
  2. Participants must have progressed within 6 months of completion of a platinum-based adjuvant, neoadjuvant, or definitive chemotherapy, or concomitant chemoradiation regimen for locally advanced disease
* Participants with non-squamous cell NSCLC of unknown epidermal growth factor receptor (EGFR) mutation status will require testing (local laboratory, or central laboratory if local testing is not available). Participants with a tumor that harbors an activating EGFR mutation will not be eligible
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry
* Estimated life expectancy of more than 12 weeks
* Adequate hematological function defined by White Blood Cell (WBC) count >= 2.5 × 10^9/L with absolute neutrophil count (ANC) >= 1.5 × 10^9/L, lymphocyte count >=0.5 × 10^9/L, platelet count >= 100 × 10^9/L, and hemoglobin >= 9 gram per deciliter (g/dL) (may have been transfused)
* Adequate hepatic function defined by a total bilirubin level less than or equal to (<=) 1.5 × the upper limit of normal (ULN) range and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels <= 2.5 × ULN for all participants
* Adequate renal function defined by an estimated creatinine clearance > 30 milliliter per minute (mL/min) according to the Cockcroft-Gault formula (or local institutional standard method).

Other protocol defined inclusion criteria could apply

Exclusion criteria

* In the United States only, participants with a squamous cell histology will be excluded
* Systemic anticancer therapy administered after disease progression during or following a platinum based combination
* Participants with non-squamous cell NSCLC whose disease harbors EGFR mutation(s) and/or anaplastic lymphoma kinase (ALK) rearrangement will not be eligible for this trial. Participants of unknown ALK and/or EGFR mutation status will require testing at screening (local laboratory, or central laboratory if local testing is not available)
* Prior therapy with any antibody/drug targeting T cell coregulatory proteins (immune checkpoints) such as PD-1, PD L1, or cytotoxic T lymphocyte antigen-4 (CTLA-4).
* Concurrent anticancer treatment
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of randomization and/or if the participant has not fully recovered from the surgery within 4 weeks of randomization
* Participants receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of the trial treatment.
* All participants with brain metastases, except those meeting the following criteria:

  1. Brain metastases have been treated locally, and
  2. No ongoing neurological symptoms that are related to the brain localization of the disease
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

  1. Participants with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
  2. Participants requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses less than or equal to (<=)10 milligram (mg) or equivalent prednisone per day
  3. Administration of steroids through a route known to result in a minimal systemic exposure are acceptable
* Previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon is acceptable as long as it is anticipated that the administration of steroids will be completed in 14 days, or that the daily dose after 14 days will be <=10 mg per day of equivalent prednisone

Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (260):
- United States (27):
  - University of Alabama, Tuscaloosa, Alabama
  - Mayo Clinic, Scottsdale , Phoenix, Arizona
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Healing Hands Oncology and Medical Care, Lawndale, California
  - Sutter Gould Medical Foundation, Modesto, California
  - Sharp Memorial Hospital, San Diego, California
  - Lynn Cancer Institute Center, Boca Raton, Florida
  - University Cancer Institute, Boynton Beach, Florida
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Florida Cancer Specialists-Broadway, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Metairie Oncologist, LLC, Metairie, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Mercy Clinic Oklahoma Communities, Inc., Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Univ. Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Center for Biomedical Research, LLC, Knoxville, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - MultiCare Health System, Tacoma, Washington
- Argentina (13):
  - Hospital Italiano Regional del Sur, Bahía Blanca
  - Clínica Universitaria Privada Reina Fabiola, Barrio General Paz
  - Centro de Oncologia e Investigacion Buenos Aires, Berazategui
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma Buenos Aires
  - CEMIC, Ciudad Autonoma Buenos Aires
  - Instituto DAMIC Fundacion Rusculleda, Córdoba
  - Centro Oncologico Riojano Integral (Cori), La Rioja
  - Centro Oncologico de Parana, Paraná
  - Hospital Universitario Austral, Pilar
  - Instituto Gamma, Rosario
  - Sanatorio Parque S.A., Rosario
  - Instituto de Oncología de Rosario, Rosario
  - Centro Medico San Roque S.R.L., San Miguel de Tucumán
- Australia (9):
  - Ballarat Base Hospital, Ballarat
  - Box Hill Hospital, Box Hill
  - Coffs Harbour Base Hospital, Coffs Harbour
  - Lyell McEwin Hospital, Elizabeth Vale
  - Greenslopes Private Hospital, Greenslopes
  - Lismore Base Hospital, Lismore
  - Royal Melbourne Hospital, Parkville
  - St John of God Hospital, Subiaco
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (6):
  - UZ Antwerpen, Edegem
  - Grand Hôpital de Charleroi, Gilly
  - UZ Leuven, Leuven
  - Centre Hospitalier de l'Ardenne, Libramont
  - C. H. U. Sart Tilman, Liège
  - AZ Delta, Roeselare
- Brazil (16):
  - Cenantron - Centro Avançado de Tratamento Oncológico S/C Ltda, Belo Horizonte
  - CEPON - Centro de Pesquisas Oncológicas de Santa Catarina, Florianópolis
  - Hospital de Caridade de Ijuí, Ijuí
  - Clínica de Neoplasias Litoral Ltda., Itajaí
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora
  - Hospital Bruno Born, Lajeado
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal
  - Oncosinos - Clínica de Oncologia - Hospital Regina, Novo Hamburgo
  - CITO - Centro Integrado de Terapia Onco-Hematológica - Hospital da Cidade de Passo Fundo, Passo Fundo
  - Hospital Mãe de Deus, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - COI - Clínicas Oncológicas Integradas, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
  - IOS - Instituto de Oncologia de Sorocaba "Dr. Gilson Delgado", Sorocaba
- Bulgaria (6):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - MHAT "Serdika", EOOD, Sofia
  - MHAT 'Tokuda Hospital Sofia', AD, Sofia
  - Shato, Ead, Sofia
  - MHAT 'Sv. Marina', EAD, Varna
- Chile (6):
  - Instituto de Terapias Oncologicas Providencia, Santiago
  - FALP - Fundación Arturo López Pérez, Santiago
  - CIEC - Centro Internacional de Estudios Clínicos, Santiago
  - Instituto Clinico Oncologico del Sur (ICOS), Temuco
  - Centro de Investigaciones Clinicas Viña del Mar, Viña del Mar
  - Hospital Clinico Viña del Mar, Viña del Mar
- Colombia (10):
  - Fundacion Cardioinfantil Instituto de Cardiologia, Bogotá
  - Instituto Nacional de Cancerologia E.S.E., Bogotá
  - Administradora Country S.A., Bogotá
  - Clinica Colsanitas S.A. sede Clinica Universitaria Colombia, Bogotá
  - Fundación Valle del Lilí, Cali
  - Centro Medico Imbanaco, Cali
  - Hemato Oncologos S.A., Cali
  - Hospital Pablo Tobón Uribe, Medellín
  - Instituto de Cancerologia S.A., Medellín
  - IPS IMAT- Instituto Medico de Alta Tecnologia - Oncomedica S.A., Montería
- Croatia (4):
  - General Hospital Dubrovnik, Dubrovnik
  - General Hospital Zadar, Zadar
  - Clinical Hospital Centar "Sestre Milosrdnice", Zagreb
  - University Clinic for Pulmonary Diseases, Zagreb
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno
  - Nemocnice Novy Jicin a.s., Nový Jičín
  - Multiscan s.r.o., Pardubice
  - Vseobecna fakultni nemocnice V Praze, Prague
  - Thomayerova nemocnice, Prague
- Denmark (2):
  - Herlev Hospital, Herlev
  - Odense Universitetshospital, Odense C
- France (11):
  - ICO - Site Paul Papin, Angers
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Hôpital Nord - AP-HM Marseille#, Marseille
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque, Pessac
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - ICO - Site René Gauducheau, Saint-Herblain
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Hungary (5):
  - Semmelweis Egyetem AOK, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Miskolci Semmelweis Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Tudogyogyintezet Torokbalint, Törökbálint
- Israel (9):
  - Assaf Harofeh Medical Center, Beer Yaakov
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Sapir Medical Center, Meir Hospital, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona
  - Ospedale Mater Salutis, Legnago (VR)
  - Ospedale Versilia, Lido di Camaiore
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Seconda Università degli Studi di Napoli, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Università Campus Bio-Medico di Roma, Roma
  - Istituto Nazionale Tumori Regina Elena IRCCS, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - Azienda Ospedaliera Ospedale Treviglio-Caravaggio di Treviglio, Treviglio
- Japan (23):
  - National Cancer Center Hospital, Chūōku
  - NHO Kyushu Cancer Center, Fukuoka
  - Osaka Prefectural Medical Center for Respiratory and Allergic Diseases, Habikino-shi
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - National Cancer Center Hospital East, Kashiwa-shi
  - Saitama Cancer Center, Kitaadachi-gun
  - Institute of Biomedical Research and Innovation Hospital, Kobe
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Kurume University Hospital, Kurume-shi
  - Miyagi Cancer Center, Natori-shi
  - Aichi Cancer Center Hospital, Okazaki-shi
  - Osaka City General Hospital, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Kinki University Hospital, Osakasayama-shi
  - Kitasato University Hospital, Sagamihara-shi
  - NHO Hokkaido Cancer Center, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Toyama University Hospital, Toyama
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama Municipal Citizen's Hospital, Yokohama
  - Kanagawa Cancer Center, Yokohama
- Mexico (8):
  - Phylasis Clinicas Research S de RL de CV, Cuautitlán Izcalli
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Fundacion Rodolfo Padilla Padilla, A.C., León
  - Health Pharma Professional Research S.A. de C.V., México
  - Winsett Rethman S.A. de C.V., Monterrey
  - Centro de Investigacion Clinica Chapultepec S.A. de C.V., Morelia
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - Centro Oncologico Estatal ISSEMyM, Toluca
- Peru (7):
  - Clinica Monte Carmelo, Arequipa
  - Hospital Nacional Almanzor Aguinaga Asenjo, Chiclayo
  - Hospital Nacional Adolfo Guevara Velasco, Cusco
  - Clinica San Borja, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
  - Clínica Ricardo Palma, Lima
  - Instituto Nacional de Enfermedades Neoplásicas, Lima
- Poland (7):
  - Szpital Specjalistyczny W Brzozowie, Podkarpacki Osrodek Onkologiczny Im.Ks.B.Markiewicza, Brzozów
  - Wojewodzkie Centrum Szpitalne Kotliny Jeleniogorskiej, Jelenia Góra
  - Samodzielny Publiczny Szpital Kliniczny nr 5 SUM, Katowice
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - SSZZOZ im. Dr Teodora Dunina w Rudce, Mrozy
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
- Romania (6):
  - Spitalul Judetean de Urgenta Alba Iulia, Alba Iulia
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris" Baia Mare, Baia Mare
  - Policlinica de Diagnostic Rapid SRL, Brasov
  - Spitalul Clinic Municipal "Dr. Gavril Curteanu" Oradea, Oradea
  - Spital Lotus SRL, Ploieşti
  - S.C Oncocenter Oncologie Clinica S.R.L, Timișoara
- Russia (6):
  - SHI "Republican Clinical Oncological Dispensary of HM RT", Kazan'
  - SHBI Moscow Clinical Scientific Center of Department of Healthcare of Moscow, Moscow
  - FSBHI Clinical research institute of phthisiopulmonology, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - St. Petersburg SHI "City Clinical Oncology Dispensary", Saint Petersburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
- Slovakia (4):
  - Nemocnica s poliklinikou Sv. Jakuba, n.o. Bardejov, Bardejov
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Ustredna vojenska nemocnica SNP Ruzomberok- Fakultna nemocnica, Ružomberok
  - Fakultna nemocnica Trnava, Trnava
- South Africa (5):
  - GVI Cape Gate Oncology Centre, Cape Town
  - GVI Rondebosch Oncology Centre, Cape Town
  - GVI Langenhoven Drive Oncology Centre, Port Elizabeth
  - University of Pretoria Oncology Department, Pretoria
  - Mary Potter Oncology Centre, Pretoria
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (15):
  - Hospital General Universitario de Alicante, Alicante
  - ICO Badalona - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario Materno-Infantil de Canarias, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon y Cajal, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital de Mataro, Mataró
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Kantonsspital Graubuenden, Chur, Switzerland
- Taiwan (6):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Turkey (Türkiye) (11):
  - Hacettepe University Medical Faculty, Ankara
  - Baskent University Ankara Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Trakya University Medical Faculty, Edirne
  - Bezmi Alem Foundation University Medical Faculty Hospital, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Fatih Universitesi Tip Fakultesi, Istanbul
  - Marmara University Pendik Research and Training Center, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medicine Faculty, Izmir
  - Konya Necmettin Erbakan University Meram Faculty of Medicine, Konya
- United Kingdom (9):
  - Royal Bournemouth General Hospital, Bournemouth
  - Bristol Haematology & Oncology Centre, Bristol
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - University College London Hospital, London
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Derriford Hospital, Plymouth
  - Mount Vernon Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- [Derived] Coon CD, Schlichting M, Zhang X. Interpreting Within-Patient Changes on the EORTC QLQ-C30 and EORTC QLQ-LC13. Patient. 2022 Nov;15(6):691-702. doi: 10.1007/s40271-022-00584-w. Epub 2022 Jun 30. PMID 35771392
- [Derived] Hrinczenko B, Iannotti N, Goel S, Spigel D, Safran H, Taylor MH, Bennouna J, Wong DJ, Kelly K, Verschraegen C, Bajars M, Manitz J, Ruisi M, Gulley JL. Long-term avelumab in advanced non-small-cell lung cancer: summaries and post hoc analyses from JAVELIN Solid Tumor. Future Oncol. 2022 Apr;18(11):1333-1342. doi: 10.2217/fon-2021-0930. Epub 2022 Feb 11. PMID 35144482
- [Derived] Park K, Ozguroglu M, Vansteenkiste J, Spigel D, Yang JC, Bajars M, Ruisi M, Manitz J, Barlesi F. Impact of subsequent immune checkpoint inhibitor treatment on overall survival with avelumab vs docetaxel in platinum-treated advanced NSCLC: Post hoc analyses from the phase 3 JAVELIN Lung 200 trial. Lung Cancer. 2021 Apr;154:92-98. doi: 10.1016/j.lungcan.2021.01.026. Epub 2021 Feb 6. PMID 33636453
- [Derived] Barlesi F, Vansteenkiste J, Spigel D, Ishii H, Garassino M, de Marinis F, Ozguroglu M, Szczesna A, Polychronis A, Uslu R, Krzakowski M, Lee JS, Calabro L, Aren Frontera O, Ellers-Lenz B, Bajars M, Ruisi M, Park K. Avelumab versus docetaxel in patients with platinum-treated advanced non-small-cell lung cancer (JAVELIN Lung 200): an open-label, randomised, phase 3 study. Lancet Oncol. 2018 Nov;19(11):1468-1479. doi: 10.1016/S1470-2045(18)30673-9. Epub 2018 Sep 24. PMID 30262187
- See also: Trial Awareness and Transparency website — http://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR100070_004
- See also: US Medical Information website, Medical Resources — http://medical.emdserono.com/en_US/home.html
- See also: Medical Information Location Map - Med Info Contacts — http://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First participant signed informed consent: 24 Mar 2015, Clinical data cut-off: 04 March 2019.
Period: Overall Study
Arm/Group | Avelumab | Docetaxel
Started | 396 | 396
Treated | 393 | 365
Completed | 393 | 365
Not Completed | 3 | 31
Not completed — Participants randomized but not treated | 3 | 31

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized to study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avelumab | Docetaxel | Total
Number analyzed (Participants) | 396 | 396 | 792
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.99) | 62.5 (9.65) | 62.7 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 123 | 250
  Male | 269 | 273 | 542
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 42 | 101
  Not Hispanic or Latino | 297 | 307 | 604
  Unknown or Not Reported | 40 | 47 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 102 | 114 | 216
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 1 | 6
  White | 273 | 262 | 535
  Not collected at the site | 14 | 14 | 28
  Other | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time in Programmed Death Ligand 1 (PD-L1) + Full Analysis Set Population (FAS)
Description: The OS time was defined as the time from randomization to the date of death. The participants who were still alive at the time of data analysis or who were lost to follow-up OS time was censored at the last recorded date that the participant was known to be alive before the data cutoff date. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from date of randomization up to 1420 days
Population: PD-L1+ FAS included all PD-L1+ tumor participants who were randomly assigned to trial treatment. The PD-L1+ participants were with greater than or equal to (>=) 1 percentage (%) of tumor cells with >=1+ positive membrane staining intensity for PD-L1 protein.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 264 | 265
months | 11.4 [9.4 to 13.8] | 10.6 [8.5 to 12.9]
Statistical Analysis 1: Comparison: Avelumab vs Docetaxel; Test type: Superiority; p = 0.0721, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.71 to 1.05]

2. Secondary Outcome: Overall Survival (OS) Time in Full Analysis Set Population
Description: as for outcome 1
Time Frame: Time from date of randomization up to 1420 days
Population: Full analysis set (FAS) included all participants who were randomized to study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 396 | 396
months | 10.6 [9.2 to 12.3] | 9.9 [8.1 to 11.9]
Statistical Analysis 1: Comparison: Avelumab vs Docetaxel; Test type: Superiority; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.77 to 1.05]

3. Secondary Outcome: Progression-Free Survival (PFS) Time in PD-L1+ Full Analysis Set Population
Description: PFS was defined as the time from date of randomization until date of the first documentation of progressive disease (PD) or death due to any cause in the absence of documented PD, whichever occurs first. PFS was assessed as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as adjudicated by independent endpoint review committee (IERC). PD was defined as at least a 20 percent (%) increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from date of randomization up to 907 days
Population: PD-L1+ FAS included all PD-L1+ tumor participants who were randomly assigned to trial treatment. The PD-L1+ participants were with >= 1 percentage of tumor cells with >=1+ positive membrane staining intensity for PD-L1 protein.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 264 | 265
months | 3.4 [2.7 to 4.9] | 4.1 [3.0 to 5.3]
Statistical Analysis 1: Comparison: Avelumab vs Docetaxel; Test type: Superiority; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.80 to 1.27]

4. Secondary Outcome: Progression-Free Survival (PFS) Time in Full Analysis Set Population
Description: as for outcome 3
Time Frame: Time from date of randomization up to 907 days
Population: Full analysis set (FAS) included all participants who were randomized to study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 396 | 396
months | 2.8 [2.7 to 3.5] | 4.2 [3.3 to 5.2]
Statistical Analysis 1: Comparison: Avelumab vs Docetaxel; Test type: Superiority; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.98 to 1.41]

5. Secondary Outcome: Number of Participants With Confirmed Best Overall Response (BOR) as Assessed by an Independent Endpoint Review Committee (IERC) in Full Analysis Set Population
Description: Confirmed BOR was determined according to RECIST v1.1 and as adjudicated by an IERC. Confirmed BOR was defined as the best response of any of the complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from the date of randomization until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. Number of participants with best overall response in each category (CR, PR, SD, PD) was reported.
Time Frame: Time from date of randomization up to 907 days
Population: Full analysis set (FAS) included all participants who were randomized to study.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 396 | 396
Participants
  Complete Response | 5 | 2
  Partial Response | 54 | 42
  Stable Disease | 129 | 158
  Non-complete Response/ Non-progressive Disease | 5 | 13
  Progressive Disease | 150 | 82
  Not Evaluable | 53 | 99

6. Secondary Outcome: Number of Participants With Confirmed Best Overall Response (BOR) as Assessed by Independent Endpoint Review Committee (IERC) in PD-L1+ Full Analysis Set Population
Description: as for outcome 5
Time Frame: Time from date of randomization up to 907 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 264 | 265
Participants
  Complete Response | 4 | 1
  Partial Response | 46 | 30
  Stable Disease | 86 | 104
  Non-complete Response/ Non-progressive Disease | 4 | 12
  Progressive Disease | 93 | 57
  Not Evaluable | 31 | 61

7. Secondary Outcome: Percentage of Participants With Objective Response as Assessed by Independent Endpoint Review Committee (IERC) in Full Analysis Set Population
Description: Percentage of participants with objective response (CR plus PR) according to RECIST v1.1 was reported. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions.
Time Frame: Time from date of randomization up to 907 days
Population: Full analysis set (FAS) included all participants who were randomized to study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 396 | 396
percentage of participants | 14.9 [11.5 to 18.8] | 11.1 [8.2 to 14.6]
Statistical Analysis 1: Comparison: Avelumab vs Docetaxel; Test type: Superiority; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.92 to 2.13]

8. Secondary Outcome: Percentage of Participants With Objective Response as Assessed by Independent Endpoint Review Committee (IERC) in PD-L1+ Full Analysis Set Population
Description: as for outcome 7
Time Frame: Time from date of randomization up to 907 days
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 264 | 265
percentage of participants | 18.9 [14.4 to 24.2] | 11.7 [8.1 to 16.2]
Statistical Analysis 1: Comparison: Avelumab vs Docetaxel; Test type: Superiority; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.08 to 2.86]

9. Secondary Outcome: Change From Baseline in European Quality of Life 5-dimensions (EQ-5D-5L) Health Outcome Questionnaire Through Composite Index Score at End of Treatment (EOT)
Description: The EQ-5D-5L health outcome questionnaire was a measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L defined health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5 items were combined to generate health profiles. These profiles were converted to a continuous single index score. The lowest possible score was -0.59 (unable to walk, unable to self-care, unable to do usual activities, extreme pain or discomfort, extreme anxiety or depression) and the highest was 1.00 (no problems in all 5 dimensions).
Time Frame: Baseline, End of treatment visit (up to Week 124)
Population: Health-related quality of life (HRQoL) analysis set was a subset of the FAS and includes all FAS participants who had 1 baseline HRQoL assessment and at least 1 post-baseline HRQoL questionnaire completed. Here, "Overall Number of Participants Analyzed" signified the participants analyzed in this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 172 | 196
units on a scale | -0.1245 (0.28021) | -0.0988 (0.26615)

10. Secondary Outcome: Change From Baseline in European Quality of Life 5-dimensions (EQ-5D-5L) Health Outcome Questionnaire Through Visual Analogue Scale (VAS) at End of Treatment (EOT)
Description: EQ-5D-5L was comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses were used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 was the worst health you can imagine and 100 was the best health you can imagine.
Time Frame: Baseline, End of treatment visit (up to Week 124)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 171 | 196
millimeter | -8.1 (22.06) | -7.0 (21.12)

11. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status at End of Treatment (EOT)
Description: EORTC QLQ-C30 was a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact). The EORTC QLQ-C30 GHS/QoL score ranged from 0 to 100; High score indicated better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Time Frame: Baseline, End of treatment visit (up to Week 124)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 172 | 196
units on a scale | -9.79 (24.506) | -9.44 (18.933)

12. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) at End of Treatment (EOT)
Description: EORTC QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The EORTC QLQ-LC13 module generated one multiple-item score assessing dyspnea and a series of single item scores assessing coughing, hemoptysis, sore mouth, dysphagia, neuropathy, alopecia, pain in chest, pain in arms or shoulder and pain in other parts. Score range: 0 (no burden of symptom domain or single symptom item) to 100 (highest burden of symptoms for symptom domains and single items).
Time Frame: Baseline, End of treatment visit (up to Week 124)
Population: Health-related quality of life (HRQoL) analysis set was a subset of the FAS and includes all FAS participants who had 1 baseline HRQoL assessment and at least 1 post-baseline HRQoL questionnaire completed. Here, "Number Analyzed" signified those participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 348 | 333
units on a scale
  Dyspnea: number analyzed (Participants) | 172 | 197
  Dyspnea | 9.95 (22.094) | 8.52 (21.285)
  Coughing: number analyzed (Participants) | 172 | 197
  Coughing | -0.58 (30.263) | -2.03 (32.582)
  Hemoptysis: number analyzed (Participants) | 172 | 197
  Hemoptysis | 0.19 (14.191) | -0.34 (16.832)
  Sore Mouth: number analyzed (Participants) | 172 | 197
  Sore Mouth | 0.78 (17.643) | 3.72 (24.920)
  Dysphagia: number analyzed (Participants) | 172 | 197
  Dysphagia | 5.62 (18.401) | 4.23 (21.538)
  Peripheral Neuropathy: number analyzed (Participants) | 172 | 197
  Peripheral Neuropathy | 0.19 (20.550) | 9.81 (30.015)
  Alopecia: number analyzed (Participants) | 172 | 197
  Alopecia | -3.10 (20.789) | 30.80 (42.582)
  Pain in Chest: number analyzed (Participants) | 172 | 197
  Pain in Chest | 4.84 (28.993) | 0.34 (26.935)
  Pain in Arm or Shoulder: number analyzed (Participants) | 172 | 197
  Pain in Arm or Shoulder | 5.62 (28.852) | 0.85 (29.439)
  Pain in Other Parts: number analyzed (Participants) | 171 | 197
  Pain in Other Parts | 8.77 (34.410) | 6.60 (30.978)

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), Drug Related Treatment Emergent Adverse Events and Treatment Emergent Adverse Events Leading to Death
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including clinically significant abnormal laboratory, vital signs and 12-lead Electrocardiogram findings), symptom, or disease temporally associated with the use of study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent events were the events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state up to 30 days after last administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Time from date of randomization up to 1420 days
Population: Safety analysis set included all participants who were administered at least 1 dose of the Investigational Medicinal Product.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 393 | 365
Participants
  TEAEs | 375 | 346
  TESAEs | 167 | 145
  Drug Related TEAEs | 252 | 313
  TEAEs Leading to Death | 64 | 51

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Severity
Description: Treatment Emergent Adverse Events were graded as per National Cancer Institute Common Terminology Criteria for Adverse Experience version 4.03 (NCI-CTCAE v 4.03). Grade 3 refers to severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care and Activity of daily living (ADL), Grade 4 refers to Life-threatening consequences; where urgent intervention indicated, Grade 5 refers to the death related to adverse event.
Time Frame: Time from date of randomization up to 1420 days
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 393 | 365
Participants
  Grade 3 or Higher | 209 | 247
  Grade 4 or Higher | 87 | 122
  Grade 5 | 63 | 51

15. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score vs. Worst Post-baseline Score
Description: ECOG performance status measured to assess participant's performance status on a scale of 0 to 5, where 0 = Fully active, able to carry on all pre-disease activities without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; 3 = Capable of only limited self-care, confined to bed/chair for more than 50 percent of waking hours; 4 = Completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5 = dead. The participants with missing worst post baseline score were also reported. ECOG performance status was reported in terms of number of participants with Baseline value vs. worst post-baseline value (i.e. highest score) combination.
Time Frame: Time from date of randomization up to 1420 days
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab | Docetaxel
Number analyzed (Participants) | 393 | 365
Participants
  Baseline score 0, worst post-baseline score 0 | 52 | 55
  Baseline score 0, worst post-baseline score 1 | 67 | 41
  Baseline score 0, worst post-baseline score 2 | 19 | 12
  Baseline score 0, worst post-baseline score 3 | 5 | 2
  Baseline score 0, worst post-baseline score 4 | 0 | 1
  Baseline score 0, worst post-baseline score 5 | 1 | 0
  Baseline score 0, worst post-baseline Missing | 0 | 6
  Baseline score 1, worst post-baseline score 0 | 6 | 1
  Baseline score 1, worst post-baseline score 1 | 157 | 172
  Baseline score 1, worst post-baseline score 2 | 47 | 41
  Baseline score 1, worst post-baseline score 3 | 23 | 8
  Baseline score 1, worst post-baseline score 4 | 3 | 2
  Baseline score 1, worst post-baseline score 5 | 1 | 1
  Baseline score 1, worst post-baseline Missing | 12 | 23

16. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) for Avelumab
Description: Serum samples were analyzed by a validated electrochemiluminesce immunoassay to detect the presence of antidrug antibodies (ADA). Samples that screened positive were subsequently tested in a confirmatory assay were tested for neutralizing antibodies (nAb). Number of participants with ADA or nAb positive results for Avelumab were reported.
Time Frame: Time from date of randomization up to 1420 days
Population: Full analysis set (FAS) included all participants who were randomized to study. Here, "Overall Number of Participants Analyzed" signified participants with at least on valid ADA result at any time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 388
Participants
  ADAs to Avelumab | 58
  NAbs to Avelumab | 14

ADVERSE EVENTS:
Time Frame: Time from date of randomization up to 1420 days.
Description: Safety analysis set included all participants who were administered at least 1 dose of the Investigational Medicinal Product.
Arm/Group | Avelumab | Docetaxel
All-Cause Mortality (participants affected / at risk) | 316/393 | 297/365
Serious Adverse Events (participants affected / at risk) | 167/393 | 145/365
Other Adverse Events (participants affected / at risk) | 320/393 | 307/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab (N=393) | Docetaxel (N=365)
Disease progression (General disorders) | 41 | 26
Asthenia (General disorders) | 6 | 3
Death (General disorders) | 6 | 4
Pain (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 3
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Sudden cardiac death (General disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia (Infections and infestations) | 9 | 19
Respiratory tract infection (Infections and infestations) | 4 | 5
Lung infection (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 2 | 2
Appendicitis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 4
Diabetic gangrene (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Klebsiella infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Meningitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 2
Peritonitis (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 5
Serratia infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 10 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Autoimmune myocarditis (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 2 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 22
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 10
Adrenal insufficiency (Endocrine disorders) | 1 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 4
Confusional state (Psychiatric disorders) | 2 | 1
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab (N=393) | Docetaxel (N=365)
Fatigue (General disorders) | 70 | 66
Asthenia (General disorders) | 55 | 64
Pyrexia (General disorders) | 50 | 33
Chills (General disorders) | 29 | 3
Oedema peripheral (General disorders) | 21 | 37
Malaise (General disorders) | 9 | 26
Mucosal inflammation (General disorders) | 5 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 77 | 46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 75 | 54
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 25 | 15
Nausea (Gastrointestinal disorders) | 56 | 57
Constipation (Gastrointestinal disorders) | 45 | 43
Diarrhoea (Gastrointestinal disorders) | 44 | 67
Vomiting (Gastrointestinal disorders) | 38 | 28
Stomatitis (Gastrointestinal disorders) | 9 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 47 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 30
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 25 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 43
Decreased appetite (Metabolism and nutrition disorders) | 79 | 76
Infusion related reaction (Injury, poisoning and procedural complications) | 56 | 8
Rash (Skin and subcutaneous tissue disorders) | 33 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 13
Weight decreased (Investigations) | 50 | 30
Neutrophil count decreased (Investigations) | 3 | 34
White blood cell count decreased (Investigations) | 2 | 21
Anaemia (Blood and lymphatic system disorders) | 50 | 81
Neutropenia (Blood and lymphatic system disorders) | 2 | 48
Headache (Nervous system disorders) | 30 | 19
Neuropathy peripheral (Nervous system disorders) | 6 | 33
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 27
Dysgeusia (Nervous system disorders) | 1 | 23
Upper respiratory tract infection (Infections and infestations) | 28 | 12
Hypothyroidism (Endocrine disorders) | 24 | 1
Insomnia (Psychiatric disorders) | 19 | 22
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT02395172/SAP_000.pdf
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT02395172/Prot_001.pdf